CLINICAL TRIAL: NCT00519532
Title: A Multicenter, Multinational, Phase 3b, Open-label Extension Trial to Evaluate the Long-term Effect of the 24-hour Transdermal Delivery of Rotigotine on Motor Function, Sleep Quality, and Nocturnal and Non-motor Symptoms in Subjects With Idiopathic Parkinson's Disease
Brief Title: Long-term Extension of RECOVER- Long-term Effect of the 24h Transdermal Delivery of Rotigotine in Subjects With Idiopathic Parkinson's Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to clinical trial supplies shortage
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP0915; EudraCT number: 2006-006907-35 (Other: EudraCT)
Record Dates: First submitted 2007-08-21; First posted 2007-08-22 (Estimated); Results first posted 2010-04-02 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2010-09

CONDITIONS: Parkinson's Disease
Keywords: Neupro®; Rotigotine; Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — rotigotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rotigotine (Experimental): Rotigotine Transdermal Patch
  Interventions: Drug: Rotigotine

INTERVENTIONS:
Drug: Rotigotine — Rotigotine transdermal patches:
  10cm2 (2mg/24h); 20cm2 (4mg/24h); 30cm2 (6mg/24h); 40cm2 (8mg/24h)
  Optimal dosing: The maximum rotigotine dose allowed is 16mg/24h
  Other Names: Neupro®

SUMMARY:
The objective of this open-label extension is to assess the long-term effect of the 24-hour transdermal delivery of rotigotine on motor function, sleep quality, and nocturnal and non-motor symptoms of Parkinson's disease. The long-term safety and tolerability of the rotigotine transdermal patch will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Completion of trial SP889

Exclusion Criteria:

* Ongoing serious adverse event assessed as related to trial medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2007-07; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (21):
- United States (2):
  - St. Petersburg, Florida
  - Salisbury, North Carolina
- Concord, Australia
- Oulu, Finland
- Germany (6):
  - Berlin
  - Dresden
  - Kassel
  - Marburg
  - Naumburg
  - Ulm
- Hungary (2):
  - Budapest
  - Nyíregyháza
- Italy (2):
  - Chieti
  - Milan
- Christchurch, New Zealand
- Olyszytn, Poland
- Cape Town, South Africa
- Spain (2):
  - Barcelona
  - Madrid
- United Kingdom (2):
  - Lancashire
  - Liverpool

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 84 subjects belong to the Enrolled Set (ES) and all of them received at least 1 dose of trial medication, so they all belong to the Safety Set (SS). 83 subjects belong to the Full Analysis Set (FAS).
Pre-assignment Details: Participant Flow information belong to the Enrolled Set (ES). Baseline Characteristics are described for the Full Analysis Set (FAS).
Period: Overall Study
Arm/Group | Rotigotine
Started | 84
Completed | 66
Not Completed | 18
Not completed — Adverse Event | 11
Not completed — Withdrawal by Subject | 5
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Rotigotine
Number analyzed (Participants) | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 34
  >=65 years | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 71
  More than one race | 0
  Unknown or Not Reported | 9
L- Dopa [Number; unit: participants]
  Early | 10
  Advanced | 73
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/ m^2] | 26.928 (4.219)
Height [Mean (Standard Deviation); unit: cm] | 170.1 (10.58)
Weight [Mean (Standard Deviation); unit: kg] | 78.3 (16.6)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in UPDRS III Score at Week 13 (End of Maintenance)
Description: The Unified Parkinson´s Disease Rating Scale Part III is an accepted and validated scale for the assessment of motor function in Parkinson´s disease. Each of the elements in the UPDRS III is measured on a scale of 0 to 4, where 0 is normal and 4 represents severe abnormalities.
  Baseline is defined as first titration visit (T1) of SP915.
Time Frame: Baseline (baseline SP915) and week 13 (End of maintenance)
Population: Full Analysis Set (FAS).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rotigotine
Number analyzed (Participants) | 76
units on a scale | -5.8 (9.4)

2. Primary Outcome: Change From Baseline in Parkinson Disease Sleep Scale (PDSS) at Week 13 (End of Maintenance)
Description: The Parkinson Disease Sleep Scale (PDSS) is a questionnaire with 15 questions to assess sleep and nocturnal disability in Parkinson´s disease. The item- scores range between 0= never and 4= very often.
  Baseline is defined as Visit 2 of previous double- blind trial SP889.
Time Frame: Baseline (baseline SP889 NCT00474058) and week 13 (End of maintenance)
Population: Full Analysis Set (FAS).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rotigotine
Number analyzed (Participants) | 78
units on a scale | -5.8 (7.8)

3. Secondary Outcome: Change From Baseline in Nocturnal Akinesia, Dystonia, and Cramps Score (NADCS) at Week 13 (End of Maintenance)
Description: Subjects were asked to assess nocturnal akinesia, dystonia and cramps, using an ordinal severity scale. While a score of 0= normal and 4= maximal severity, subjects could also rate their symptoms with values of 0.5, 1.5, 2.5, 3.5. The nocturnal akinesia score was used to evaluate motor performance while the dystonia and cramps scores were used to evaluate sleep.
  Baseline is defined as Visit 2 of previous double- blind trial SP889.
Time Frame: Baseline (baseline SP889 NCT00474058) and week 13 (End of maintenance)
Population: Full Analysis Set (FAS).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rotigotine
Number analyzed (Participants) | 79
units on a scale | -1.5 (2.1)

4. Secondary Outcome: Change From Baseline in Number of Nocturias at Week 13 (End of Maintenance)
Description: The change in number of nocturias was used to evaluate improvements in sleep disorders.
  Baseline is defined as Visit 2 of previous double- blind trial SP889.
Time Frame: Baseline (baseline SP889 NCT00474058) and week 13 (End of maintenance)
Population: Full Analysis Set (FAS).
Measure: Mean (Standard Deviation); unit: Nocturias
Arm/Group | Rotigotine
Number analyzed (Participants) | 78
Nocturias | -0.4 (1.2)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected over the whole trial period from Visit 1 to the Safety Follow- Up Visit.
Description: Serious and non- serious Adverse Events (AEs) refer to the Safety Set (SS). The SS includes all subjects who received at least 1 dose of trial medication.
Arm/Group | Rotigotine
Serious Adverse Events (participants affected / at risk) | 16/84
Other Adverse Events (participants affected / at risk) | 55/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotigotine (N=84)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Atrioventricular block third degree (Cardiac disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Reflux oesophagitis (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Application site vesicles (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Death (General disorders) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 (3)
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 (1)
Eosinophil count increased (Investigations) | 1 (1)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Syncope vasovagal (Nervous system disorders) | 1 (1)
Peroneal nerve palsy (Nervous system disorders) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotigotine (N=84)
Nausea (Gastrointestinal disorders) | 10 (13)
Vomiting (Gastrointestinal disorders) | 5 (6)
Constipation (Gastrointestinal disorders) | 5 (6)
Application site pruritus (General disorders) | 8 (10)
Application site erythema (General disorders) | 10 (12)
Application site irritation (General disorders) | 5 (6)
Oedema peripheral (General disorders) | 8 (10)
Urinary tract infection (Infections and infestations) | 7 (8)
Nasopharyngitis (Infections and infestations) | 5 (6)
Fall (Injury, poisoning and procedural complications) | 10 (11)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6)
Dyskinesia (Nervous system disorders) | 9 (9)
Parkinson´s disease (Nervous system disorders) | 8 (11)
Dizziness (Nervous system disorders) | 9 (11)
Somnolence (Nervous system disorders) | 11 (12)
Headache (Nervous system disorders) | 5 (11)
Hallucination (Psychiatric disorders) | 11 (22)
Insomnia (Psychiatric disorders) | 7 (7)

LIMITATIONS AND CAVEATS:
Because the manufacturing process for rotigotine patches was changed, enrollment into SP915 was stopped in April 2008 to ensure sufficient trial medication for all subjects enrolled at that time to complete the trial according to the protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that is confidential and compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.